CLINICAL TRIAL: NCT03365726
Title: Intraoperative Stress Test With Dobutamine and Speckle Tracking to Decrease Postoperative Mortality
Brief Title: Intraoperative Dobutamine Stress Test With Speckle Tracking to Decrease Postoperative Mortality (ISTMO)
Acronym: ISTMO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Collaborators: A.O. Ospedale Papa Giovanni XXIII (Other); Centre de Recherche de l'Institut Universitaire de Cardiologie et de Pneumologie de Quebec (Other)
Responsible Party: Principal Investigator, Lina Pietropaoli, MD, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 15-228-MUHC
Record Dates: First submitted 2017-11-22; First posted 2017-12-07 (Actual); Last update posted 2018-03-19 (Actual); Status verified 2018-03

CONDITIONS: Mortality After Major Non Cardiac Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DST (dobutamine-stress-test) (Experimental): dobutamine stress echocardiography performed to patients undergoing major surgery
  Interventions: Diagnostic Test: Dobutamine stress test with trans-esophageal echocardiography
- NDST (no-dobutamine-stress-test) (No Intervention): patients refused the dobutamine stress test and transesophageal echocardiography measured the troponin level in first 24 hours after surgery

INTERVENTIONS:
Diagnostic Test: Dobutamine stress test with trans-esophageal echocardiography — Dobutamine stress echocardiography will be performed: before skin incision and at the end of surgery.
  After a TEE evaluation at rest to assess myocardial structure, function and potential regional wall motion abnormalities, dobutamine infusion will be started
  * If no regional wall motion abnormalities will be detected, a dobutamine stress echocardiography will be started at the range infusion of 50 γ/kg/min (ADST: Accelerated Dobutamine Stress Test). The Test will be continued up to the 85% of maximum heart rate adjusted for the patient age and echo images will be stored.
  * If regional wall motion abnormalities are present, a gradual dobutamine stress test will be started at the initial dose of 10 mcg/kg/min (GDST: Gradual Dobutamine Stress Test) and it will be increased every 3 minutes until the 85% of maximum heart rate, adjusted for patient's age (maximal dose: 40 mcg/kg/min) and echo images will be stored.
  Arms: DST (dobutamine-stress-test)

SUMMARY:
Perioperative adverse cardiovascular events are the leading cause of morbidity and mortality after noncardiac surgery. The implications of perioperative cardiac complications on morbidity and mortality, in-hospital and long-term care, and resource utilization are enormous. The continuously increasing proportion of elderly patients presenting for noncardiac surgery raises serious concerns regarding adverse cardiac events in the perioperative period. The responsibility for early diagnosis and prompt treatment of cardiac complications during surgery rests squarely with the anesthesiologist. Reliable intraoperative identification of patients at high risk for postoperative AMI and/or death is currently inadequate, but may confer substantial benefits to patients as preventive measures could be instituted. A reliable and reproducible quantitative measure of regional and global myocardial function could improve preoperative risk stratification and guide anesthetic management when acute changes in myocardial function occur.

In the present study is hypothesized that intraoperative dobutamine stress echocardiography by 2-dimensional speckle tracking echocardiography can identify patients at higher risk of perioperative adverse cardiac events.

ELIGIBILITY:
Inclusion Criteria:

* Any laparotomy
* Any thoracotomy
* Any hip surgery
* Any complex oncologic surgery o Any thoracoscopy

Exclusion Criteria:

* Females older than 80 year old
* Patients on chronic systemic corticosteroid therapy
* Diagnosed pharyngeal or gastro-esophageal pathologies (such as esophageal varices, stricture, diverticula, tumor, esophagitis, Mallory- Weiss tear, or previous surgery for any of these)
* Signs and symptoms of severe pharyngeal or gastro-esophageal pathologies (including odynophagia, dysphagia)
* Emergency surgery
* Age less than 50 year old

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 2016-01-19 (Actual); Primary Completion 2018-01-19 (Actual); Study Completion 2019-01-19 (Estimated)

PRIMARY OUTCOMES:
mortality | 30 days
  mortality

SECONDARY OUTCOMES:
myocardial infarction | within 30 days after surgery
  new ECG changes with troponin increase

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Donatelli, MD, Principal Investigator — MUHC - McGill University Health Centre; Ferdinando Luca Lorini, MD, Principal Investigator — Ospedale Papa Giovanni XXIII; Lina Pietropaoli, MD, Study Director — MUHC - McGill University Health Centre
Locations (1):
- MUHC, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vascular Events In Noncardiac Surgery Patients Cohort Evaluation (VISION) Study Investigators; Devereaux PJ, Chan MT, Alonso-Coello P, Walsh M, Berwanger O, Villar JC, Wang CY, Garutti RI, Jacka MJ, Sigamani A, Srinathan S, Biccard BM, Chow CK, Abraham V, Tiboni M, Pettit S, Szczeklik W, Lurati Buse G, Botto F, Guyatt G, Heels-Ansdell D, Sessler DI, Thorlund K, Garg AX, Mrkobrada M, Thomas S, Rodseth RN, Pearse RM, Thabane L, McQueen MJ, VanHelder T, Bhandari M, Bosch J, Kurz A, Polanczyk C, Malaga G, Nagele P, Le Manach Y, Leuwer M, Yusuf S. Association between postoperative troponin levels and 30-day mortality among patients undergoing noncardiac surgery. JAMA. 2012 Jun 6;307(21):2295-304. doi: 10.1001/jama.2012.5502. PMID 22706835
- [Background] Devereaux PJ, Xavier D, Pogue J, Guyatt G, Sigamani A, Garutti I, Leslie K, Rao-Melacini P, Chrolavicius S, Yang H, Macdonald C, Avezum A, Lanthier L, Hu W, Yusuf S; POISE (PeriOperative ISchemic Evaluation) Investigators. Characteristics and short-term prognosis of perioperative myocardial infarction in patients undergoing noncardiac surgery: a cohort study. Ann Intern Med. 2011 Apr 19;154(8):523-8. doi: 10.7326/0003-4819-154-8-201104190-00003. PMID 21502650
- [Background] Landesberg G, Beattie WS, Mosseri M, Jaffe AS, Alpert JS. Perioperative myocardial infarction. Circulation. 2009 Jun 9;119(22):2936-44. doi: 10.1161/CIRCULATIONAHA.108.828228. No abstract available. PMID 19506125
- [Background] Pearse RM, Moreno RP, Bauer P, Pelosi P, Metnitz P, Spies C, Vallet B, Vincent JL, Hoeft A, Rhodes A; European Surgical Outcomes Study (EuSOS) group for the Trials groups of the European Society of Intensive Care Medicine and the European Society of Anaesthesiology. Mortality after surgery in Europe: a 7 day cohort study. Lancet. 2012 Sep 22;380(9847):1059-65. doi: 10.1016/S0140-6736(12)61148-9. PMID 22998715
- [Background] Rose J, Weiser TG, Hider P, Wilson L, Gruen RL, Bickler SW. Estimated need for surgery worldwide based on prevalence of diseases: a modelling strategy for the WHO Global Health Estimate. Lancet Glob Health. 2015 Apr 27;3 Suppl 2(Suppl 2):S13-20. doi: 10.1016/S2214-109X(15)70087-2. PMID 25926315
- [Background] Weiser TG, Regenbogen SE, Thompson KD, Haynes AB, Lipsitz SR, Berry WR, Gawande AA. An estimation of the global volume of surgery: a modelling strategy based on available data. Lancet. 2008 Jul 12;372(9633):139-144. doi: 10.1016/S0140-6736(08)60878-8. Epub 2008 Jun 24. PMID 18582931
- [Background] Garutti I, Paniagua P, Cruz P, Maestre ML, Fernandez-Riveira C, Alonso-Coello P; Spanish VISION Investigators. Analytic comments of the initial results of the VISION (Vascular events In noncardiac Surgery patIents cOhort evaluatioN): Association between troponin T and mortality at 30 days in noncardiac surgery patients. Rev Esp Anestesiol Reanim. 2013 Jun-Jul;60(6):304-7. doi: 10.1016/j.redar.2012.10.015. Epub 2012 Dec 20. No abstract available. PMID 23261223
- [Background] Hoffmann R, Marwick TH, Poldermans D, Lethen H, Ciani R, van der Meer P, Tries HP, Gianfagna P, Fioretti P, Bax JJ, Katz MA, Erbel R, Hanrath P. Refinements in stress echocardiographic techniques improve inter-institutional agreement in interpretation of dobutamine stress echocardiograms. Eur Heart J. 2002 May;23(10):821-9. doi: 10.1053/euhj.2001.2968. PMID 12009723
- [Background] Moonen M, Lancellotti P, Zacharakis D, Pierard L. The value of 2D strain imaging during stress testing. Echocardiography. 2009 Mar;26(3):307-14. doi: 10.1111/j.1540-8175.2008.00864.x. PMID 19291016
- [Background] Amundsen BH, Helle-Valle T, Edvardsen T, Torp H, Crosby J, Lyseggen E, Stoylen A, Ihlen H, Lima JA, Smiseth OA, Slordahl SA. Noninvasive myocardial strain measurement by speckle tracking echocardiography: validation against sonomicrometry and tagged magnetic resonance imaging. J Am Coll Cardiol. 2006 Feb 21;47(4):789-93. doi: 10.1016/j.jacc.2005.10.040. Epub 2006 Jan 26. PMID 16487846
- [Background] Cho GY, Chan J, Leano R, Strudwick M, Marwick TH. Comparison of two-dimensional speckle and tissue velocity based strain and validation with harmonic phase magnetic resonance imaging. Am J Cardiol. 2006 Jun 1;97(11):1661-6. doi: 10.1016/j.amjcard.2005.12.063. Epub 2006 Apr 19. PMID 16728234
- [Background] Aggeli C, Lagoudakou S, Felekos I, Panagopoulou V, Kastellanos S, Toutouzas K, Roussakis G, Tousoulis D. Two-dimensional speckle tracking for the assessment of coronary artery disease during dobutamine stress echo: clinical tool or merely research method. Cardiovasc Ultrasound. 2015 Oct 24;13:43. doi: 10.1186/s12947-015-0038-z. PMID 26498476
- [Background] Reant P, Labrousse L, Lafitte S, Bordachar P, Pillois X, Tariosse L, Bonoron-Adele S, Padois P, Deville C, Roudaut R, Dos Santos P. Experimental validation of circumferential, longitudinal, and radial 2-dimensional strain during dobutamine stress echocardiography in ischemic conditions. J Am Coll Cardiol. 2008 Jan 15;51(2):149-57. doi: 10.1016/j.jacc.2007.07.088. PMID 18191740
- [Background] Yu Y, Villarraga HR, Saleh HK, Cha SS, Pellikka PA. Can ischemia and dyssynchrony be detected during early stages of dobutamine stress echocardiography by 2-dimensional speckle tracking echocardiography? Int J Cardiovasc Imaging. 2013 Jan;29(1):95-102. doi: 10.1007/s10554-012-0074-9. Epub 2012 May 25. PMID 22628053
- [Background] Pellikka PA, Nagueh SF, Elhendy AA, Kuehl CA, Sawada SG; American Society of Echocardiography. American Society of Echocardiography recommendations for performance, interpretation, and application of stress echocardiography. J Am Soc Echocardiogr. 2007 Sep;20(9):1021-41. doi: 10.1016/j.echo.2007.07.003. No abstract available. PMID 17765820
- [Background] Lang RM, Bierig M, Devereux RB, Flachskampf FA, Foster E, Pellikka PA, Picard MH, Roman MJ, Seward J, Shanewise JS, Solomon SD, Spencer KT, Sutton MS, Stewart WJ; Chamber Quantification Writing Group; American Society of Echocardiography's Guidelines and Standards Committee; European Association of Echocardiography. Recommendations for chamber quantification: a report from the American Society of Echocardiography's Guidelines and Standards Committee and the Chamber Quantification Writing Group, developed in conjunction with the European Association of Echocardiography, a branch of the European Society of Cardiology. J Am Soc Echocardiogr. 2005 Dec;18(12):1440-63. doi: 10.1016/j.echo.2005.10.005. No abstract available. PMID 16376782
- [Background] Wu WC, Schifftner TL, Henderson WG, Eaton CB, Poses RM, Uttley G, Sharma SC, Vezeridis M, Khuri SF, Friedmann PD. Preoperative hematocrit levels and postoperative outcomes in older patients undergoing noncardiac surgery. JAMA. 2007 Jun 13;297(22):2481-8. doi: 10.1001/jama.297.22.2481. PMID 17565082